CLINICAL TRIAL: NCT02403908
Title: Catheter Denervation of Pulmonary Arteries in The Treatment of Idiopathic (PAH) & Secondary Pulmonary Hypertension (PH)
Brief Title: Catheter Denervation of Pulmonary Arteries in Treatment of IPAH & SPAH
Acronym: CADOPA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Aleksander Ernst, Professor if Internal Medicine & Cardiology, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRZZ-2014 Project Number:2505
Record Dates: First submitted 2015-03-11; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Hypertension, Pulmonary
Keywords: radiofrequency denervation, pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PADN groups (radiofrequency denervation) (Experimental): An 8-F long sheath will be inserted through the femoral vein and advanced to the main PA (MPA). The nMARQ Circular or Crescent (Biosense Webster) catheter will be advanced along this long sheath. After gently withdrawing the sheath and pushing the PADN catheter, the tip will be released from the sheath. Then, the tip of the catheter will be positioned first at the ostium of the left PA (Level 1 of ablation, <2 mm distal to orifice. After ablation at this level, the catheter tip will be positioned at the ostium of right PA (Level 2 of ablation, <2mm proximal to the bifurcation level). Finally, denervation of main pulmonary artery will be done by pulling the denervation catheter back into Level 3 of ablation (<2 mm proximal to both ostia of right and left PA-s) into main pulmonary artery.
  Interventions: Device: nMARQ Circular and Crescent catheters
- SHAM group (No Intervention): non-treated patients (controls)

INTERVENTIONS:
Device: nMARQ Circular and Crescent catheters — Radiofrequency denervation of right and left pulmonary arteries ostia and of main pulmonary artery <2 mm proximal from both ostia of right and left pulmonary arteries.
  Other Names: Radiofrequency denervation
  Arms: PADN groups (radiofrequency denervation)

SUMMARY:
The aim of research proposal is to assess and compare the safety and efficacy of radiofrequency denervation of pulmonary arteries on decrease in pulmonary vascular resistance and mean pulmonary artery pressure (MPAP) in 20 patients with IPAH (mean pulmonary artery pressure >25 mmHg) and in 20 patients with secondary pulmonary hypertension due to pulmonary disease or due to left heart disease not responding optimally to medical therapy.

DETAILED DESCRIPTION:
METHODS:

Patient population. Patients with IPAH and SPAH (defined as a mean PAP >25 mm Hg at rest) not responding optimally to current medical therapy (defined as a reduction of <5mmHg in the resting mean PAP during medication, or unchanged 6-min walk test (6MWT) defined as increment of 6MW distance <50 m) will be eligible for the study. The patients will be informed that they have the right to withdraw their informed consent at any time. After signing a previously approved institutional written informed consent 20 patients with proven IPAH and 20 patients with proven SPAH and 20 control patients (10 with IPAH and 10 with SPAH) will be randomly assigned to radiofrequency denervation of pulmonary arteries or to sham group. Patients of age <18 years, patients with structural heart diseases with left-to right shunting and/or with Eisenmenger syndrome will be excluded from the trial. Medical treatment before enrollment including a diuretics sildenafil or bosentan or digoxin or any other necessary medication will not be discontinued. Blood samples will be obtained for N-terminal brain natriuretic peptide (NT-BNP), troponin T, mbCK, CK and other usually accepted biological markers of pulmonary hypertension levels before, immediately after the pulmonary artery denervation (PADN) procedure, and at 3 and 6 months following the PADN procedure. For the assessment of potential anatomical complications at the sight of PADN a multisliced computed tomography angiography of pulmonary trunk and pulmonary arteries will be obtained before and 6 months after PADN procedure. Assessment of functional capacity (9) will be determined by the six-minutes walk test (6MWT), followed by an assessment of dyspnea using the Borg scale (10). The 6MWT will be performed at 3 month and 6 months following the PADN procedure. The World Health Organization classification (11) at rest and during exercise will be recorded by a physician blinded to the study design.

Echocardiography will be performed at 3 month and 6 months following the procedure. Echocardiographic studies will be done using a Vivid 7 ultrasound system with a standard imaging transducer (General Electric Co., Easton Turnpike, Connecticut). All of the measurements will be performed according the recommendations of the American Society of Echocardiography (12). Digital echocardiographic data that contained a minimum of 3 consecutive beats (or 5 beats in cases of atrial fibrillation) will be acquired and analyzed. Right ventricular (RV) systolic pressure is equal to systolic PAP in the absence of pulmonary stenosis. Systolic PAP is equal to the sum of the right atrial (RA) pressure and the RV-to-RA pressure gradient during systole. RA pressure will be estimated based on the echocardiographic features of the inferior vena cava and assigned a standard value (13). The RV-to-RA pressure gradient will be calculated as 4vt2 using the modified Bernoulli equation, where vt is the velocity of the tricuspid regurgitation jet in m/s. The mean PAP will be estimated according to the velocity of the pulmonary regurgitation jet in m/s. The tricuspid excursion index (Tei) (14) is defined as (A-B)/B, where A is the time interval between the end and the onset of tricuspid annular diastolic velocity, and B is the duration of tricuspid annular systolic velocity (or the RV ejection time). PA compliance for patients will be calculated as the stroke volume divided by pulse pressure (systolic PAP minus diastolic PAP). Hemodynamic measurements and blood oxygen pressure/saturation determinations from the RA, RV, and PA will be performed as previously described using right heart catheterization before and immediately after the PADN procedure. These measurements will be repeated at 24 h, 3 months and 12 months. Measurements of resting RA pressure, RV pressure, systolic/diastolic/mean PAP, PA occlusive pressure (PAOP), cardiac output (CO) and mixed venous oxygen saturation will be recorded. The pulmonary vascular resistance (PVR) [PVR ¼(mean PAP- PAOP)/CO] and transpulmonary pressure gradient (TPG ¼ mean PAP- PAOP) will then be calculated. All of the measurements will be recorded at the end of expiration. Five criteria (15-17) will be used to evaluate whether a PAOP measurement was valid: 1) the PAOP was less than the diastolic PAP; 2) the tracing was comparable to the atrial pressure waveform; 3) the fluoroscopic image exhibited a stationary catheter following inflation; 4) free flow was present within the catheter (flush test); and 5) highly oxygenated blood (capillary) was obtained from the distal portion in the occlusion position. If the PAOP measurement was unreliable, the left ventricular end-diastolic pressure will then be measured and used rather than the PAOP.

The blood samples from the superior vena cava and PA will be obtained for the measurements of oxygen pressure and saturation. PADN procedure. A baseline PA angiography will be performed to identify the PA bifurcation level and calculate the PA diameter. An 8-F long sheath will be inserted through the femoral vein and advanced to the main PA (MPA). The PADN catheter will be advanced along this long sheath. After gently withdrawing the sheath and pushing the PADN catheter, the tip will be released from the sheath. Then, by slightly rotating and pushing the handle the tip will be positioned first at the ostium of the left PA (Level 1 of ablation, <2 mm distal to orifice. After ablation at this level, the catheter tip will be positioned at the ostium of right PA (Level 2 of ablation, <2mm proximal to the bifurcation level). Finally, denervation of main pulmonary artery will be done by pulling the denervation catheter back into Level 3 of ablation (<2 mm proximal to both ostia of right and left PA-s) into main pulmonary artery.Three criteria will be used to ensure that the electrodes were tightly in contact with the endovascular surface: 1) strong manual resistance when rotating the handle; 2) inability to advance distally or ease in, withdrawing proximally 3) angiographic confirmation and 4) actual electrode contact pressure (gm) readings provided by RF denervation system used. The procedure will be stopped if the patient complained of intolerable chest pain. The electrocardiogram and hemodynamic pressure will be monitored and continuously recorded throughout the procedure. Procedural success will be defined as a reduction in the mean PAP >10 mm Hg (as measured by the Swan-Ganz catheter), and there were no complications. The patients will be monitored in the intensive cardiac care unit for at least 24 h after the PADN procedure. Commercially available and approved radiofrequency technology for pulmonary vein isolation will be utilized for new clinical indication.

Peri-procedural medications. An intravenous bolus of 5,000 U of unfractionated heparin will be given immediately following the insertion of the venous sheath. An additional approximately 2,000 to 3,000 U of heparin will be added if the procedural time exceeds 1 h. Following the procedure, oral warfarin will be prescribed and adjusted according to the international normalized ratio to be between 2 and 2.5 for all patients. If there would be contraindications for warfarin, aspirin (100 mg/day) and clopidogrel (75 mg/day) will be prescribed indefinitely. Immediately after the PADN procedure, all medications (diuretics, sildenafil, bosentan, beraprost, digoxin etc.) will be discontinued for 24h.

Endpoints. The primary endpoints will be decrease in mean PAP and pulmonary vascular resistance at 3 and 6 months and improvement of functional capacity by the 6MWT. Clinical adverse events (including PA perforation/dissection, acute thrombus formation in the PA, all-cause death, rehospitalization due to PAH, and lung transplantation) will be secondary endpoints and will be assessed by an independent event committee. Statistical analysis. Continuous variables will be expressed as mean + SD. Differences in continuous variables between different time points in the PADN group will be analyzed using paired-sample Student t tests or Wilcoxon signed- rank sum tests, as appropriate nonparametric statistical methods. Each patient in the trial will serve as his/her own control before and after PADN and sham group patients as a control group of overall efficacy of the procedure. The categorical variables will be compared using the Fisher exact test. Statistical significance will be defined as a 2-sided p value < 0.05. All of the analyses will be performed using WinStat statistical software package for Microsoft Excel, version 2009.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IPAH and SPAH (defined as a mean PAP >25 mm Hg at rest) not responding optimally to current medical therapy (defined as a reduction of <5mmHg in the resting mean PAP during medication, or unchanged 6-min walk test (6MWT) defined as increment of 6MW distance <50 m) will be eligible for the study.

Exclusion Criteria:

- Patients of age <18 years, patients with structural heart diseases with left-to right shunting and/or with Eisenmenger syndrome will be excluded from the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
decrease in mean PAP | immeditely after PADN, and three and six months after PADN
decrease in pulmonary vascular resistance | immeditely after PADN, and three and six months after PADN
improvement of functional capacity by the 6MWT. | 48 hours after PADN, and three and six months after PADN

SECONDARY OUTCOMES:
Major clinical adverse events (MACE) including PA perforation/dissection, acute thrombus formation in the PA, all-cause death, MI, stroke | immediately after PADN, and three and six months after PADN

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital centre Zagreb, Zagreb, Croatia